CLINICAL TRIAL: NCT05244811
Title: Treatment of Functional Ovarian Cyst Randomised Clinical Trial
Brief Title: Treat of Functional Ovarian Cysts by Compare Between Cocs and Progesterone Only Pills
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelhamed Khaled Abdelhameed Farghal, resident doctor in gynaecology and obstetric department in nasser general hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ovarian cysts
Record Dates: First submitted 2022-01-09; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Contraceptives, Oral, Combined; Progestins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- use of placebo in treatment of functional ovarian cyst (Placebo Comparator): trial the effect of placebo in treatment of functional ovarian cyst
  Interventions: Drug: Combined Oral Contraceptive; Drug: Progestin
- use of cocs in treatment of functional ovarian cyst (Active Comparator): trial of the effectiveness of cocs in the treatment of functional ovarian cyst
  Interventions: Drug: Combined Oral Contraceptive; Drug: Progestin
- use of progesterone in treatment of functional ovarian cyst (Active Comparator): comparison between the effect of progesterone in the treatment of functional ovarian cyst with the effect of cocs
  Interventions: Drug: Combined Oral Contraceptive; Drug: Progestin

INTERVENTIONS:
Drug: Combined Oral Contraceptive — effect of cocs in treatment of ovarian cysts
  Other Names: cyclo progynova
Drug: Progestin — effect of progestin in treatment of ovarian cystn
  Other Names: primalot-nor

SUMMARY:
comparison between cocs and progesterone only containing pills in treatment of fuctional ovarian cyst

DETAILED DESCRIPTION:
Ovarian cyst is a blister-like sac, which is formed on the surface of ovary during or after ovulation . Most of them are made in reproductive age and are harmless ; these cysts do not cause any symptom and are resolved without treatment , but sometimes they cause health problems that require special attention, and even may lead to infertility. Normal function of ovary is the periodic release of ovums and the production of the steroid hormones of estradiol and progesterone . Both activities are integrated in the continuous repetitive process of follicle maturation, ovulation, and corpus luteum formation and regression. Mature follicle is ruptured and releases ovum during ovulation and corpus luteum is produced from empty follicle if pregnancy does not occur corpus luteum is regressed, due to the absence of hCG (human chorionic gonadotropin). Sometimes this procedure does not happen normally, which results in the formation of ovarian cysts Therefore, functional ovarian cysts are different from ovarian growths induced by other pathological problems most of them regress spontaneously in two or three cycles , but if a cyst gets large, it can twist, be ruptured, or bleed and become very painful .

A functional type of ovarian cyst forms because of slight changes in the way of making or releasing an ovum by the ovary . There are two types of such cysts:

1. The follicular cyst, which occurs when the sac on ovary does not release an egg and the sac swells up with fluid
2. The luteal cyst, which is formed when the sac releases an egg and then reseals and fills with fluid

Most functional ovarian cysts are asymptomatic , the larger the cyst, the more likely the symptom. The symptoms are pain or aching in lower abdomen, menstrual irregularity, vaginal bleeding, dyspareunia, etc.; sometimes the cyst is ruptured and causes peritoneal irritation with presentations such as nausea and vomiting or sudden onset of pain, hemorrhagic cyst, intra-abdominal bleeding, and emergency conditions . Some other manifestations such as nausea and vomiting may be felt before the occurrence of such events . Regular pelvic examination is recommended for some patients with the history of such cysts; they also may need regular sonography . Oral contraceptive pills (OCPs) are prescribed by some physician to shrink the cyst, if it is persistent and makes discomfort . Although it seems that they are not effective enough compared with close observation, and even some researchers reported no benefits for OCPs, some others prescribed them before any surgical practices ; therefore, the current study aimed at evaluating this issue. For this purpose, some patients who referred to a private clinic were selected in order to compare the effect of OCPs with close observation in the clinical management of functional ovarian cysts. dyspareunia, or the cysts may be found accidentally on voluntary sonography without any symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The current randomized, clinical trial was performed on females with:-

  1. functional ovarian cysts (4 to 8 cm in diameter)
  2. in reproductive age, within the age range of 18 to 48 years, referred to the Clinic of Gynecological Diseases in a private hospital as outpatient The cysts were identified by transvaginal ultrasonography

Exclusion Criteria:

* were history of:-

  1. endometrioma.
  2. Other non-functional .ovarian neoplasm
  3. OCPs consumption during the last three months The patients were randomly divided into three equals

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
treatment of functional ovarian cysts | one year
  rate of treatment of combined oral contraceptive pills in functional ovarian cyst compared with cases who will receive progesterone only pills

REFERENCES:
- [Background] Formuso C, Stracquadanio M, Ciotta L. Myo-inositol vs. D-chiro inositol in PCOS treatment. Minerva Ginecol. 2015 Aug;67(4):321-5. Epub 2015 Feb 11. PMID 25670222
- [Background] Wu XK, Stener-Victorin E, Kuang HY, Ma HL, Gao JS, Xie LZ, Hou LH, Hu ZX, Shao XG, Ge J, Zhang JF, Xue HY, Xu XF, Liang RN, Ma HX, Yang HW, Li WL, Huang DM, Sun Y, Hao CF, Du SM, Yang ZW, Wang X, Yan Y, Chen XH, Fu P, Ding CF, Gao YQ, Zhou ZM, Wang CC, Wu TX, Liu JP, Ng EHY, Legro RS, Zhang H; PCOSAct Study Group. Effect of Acupuncture and Clomiphene in Chinese Women With Polycystic Ovary Syndrome: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2502-2514. doi: 10.1001/jama.2017.7217. PMID 28655015